CLINICAL TRIAL: NCT01203306
Title: Phase II Study of the Combination of Bevacizumab Plus Somatostatin Analogue and Metronomic Capecitabine in Patients With Advanced Inoperable Well-Differentiated Neuroendocrine Tumors
Brief Title: Bevacizumab Plus Somatostatin Analogue and Metronomic Capecitabine in Patients With Advanced Neuroendocrine Tumors
Acronym: XELBEVOCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Alfredo Berruti, Dipartimento di Scienze Cliniche e Biologiche - Università di Torino
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2006-004748-22
Record Dates: First submitted 2010-09-09; First posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-07

CONDITIONS: Neuroendocrine Carcinomas
Keywords: bevacizumab; somatostatin analogue; metronomic capecitabine; neuroendocrine tumors
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors | interventions — Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drugs: bevacizumab + octreotide LAR + capecitabine (Experimental): bevacizumab + octreotide + metronomic capecitabine
  Interventions: Drug: bevacizumab + octreotide LAR + capecitabine

INTERVENTIONS:
Drug: bevacizumab + octreotide LAR + capecitabine — long acting octreotide acetate at a dose of 20 or 30 mg administered intramuscularly every 4 weeks; Bevacizumab at a dose of 5 mg/kg every 2 weeks; orally capecitabine administered at a dose of 2000 mg/daily
  Other Names: Avastin; Sandostatin LAR; Xeloda

SUMMARY:
Well differentiated neuroendocrine (NE) carcinomas have low proliferative activity and conventional chemotherapy is not recommended. Metronomic chemotherapy, i.e. the frequent administration of cytotoxic drugs at low doses, has demonstrated antiangiogenetic properties. Since well differentiated NE carcinomas are highly vascular, there is a rationale for testing metronomic chemotherapy and antiangiogenetic drugs. This is a national, multicenter, phase II study.

DETAILED DESCRIPTION:
Metastatic or locally advanced well differentiated neuroendocrine carcinoma will be treated with a combination of bevacizumab (5 mg/kg) plus octreotide LAR (long- acting release) 20/30 mg plus capecitabine administered on a metronomic schedule (2000 mg/day).

Patients with stable disease, complete or partial response will continue treatment until progressive disease or unacceptable toxicity.

Primary endpoint: the response to treatment, evaluated according to the RECIST criteria.

Secondary endpoint: - toxicity, graded according to the NCI-CTG criteria;

* symptomatic response: evaluated according to the changes in both the frequency and intensity of symptoms;
* biochemical response: evaluated considering the changes in the tumor marker levels (circulating Chromogranin A);
* relationship between vascular endothelial growth factor (VEGF) polymorphisms and response to treatment;
* time to progression and survival: measured from the date of treatment start to the date of progression and the date of last follow-up or death, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosis of well-differentiated neuroendocrine carcinoma
* Inoperable disease
* Age > 18
* ECOG Performance Status 0-2
* Life expectancy of at least 12 weeks
* Measurable and/or evaluable lesions according to RECIST criteria
* Radiological documentation of disease progression
* Adequate bone marrow reserve
* Adequate hepatic and renal function
* Urine dipstick of proteinuria < 2+
* Written informed consent
* Comply with the protocol procedures

Exclusion criteria:

* Serious non-healing wound or ulcer
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled hypertension
* Clinically significant cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Current or recent ongoing treatment with anticoagulants for therapeutic purposes
* Chronic, daily treatment with high-dose aspirin (>325 mg/day) or other medications known to predispose to gastrointestinal ulceration
* Patients with severe renal impairment (creatinine clearance below 30 ml/min)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-05 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
time to progression | 36 months

SECONDARY OUTCOMES:
Toxicity | two years
  All adverse events encountered during the clinical study will be reported. The intensity of clinical adverse events will be graded according to the NCI Common Toxicity Criteria (CTC) version 3.0 grading system.
Time to Treatment Failure (TTF) | two years
  TTF is the time from first day of treatment to the first occurrence of any adverse events with withdrew prematurely the treatment.
Overall survival (OS) | 48 months
  Overall survival (OS) will be computed as the time between the first day of treatment and the date of death or the last date the patient was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, MD, PhD, Study Director — Medical Oncology, Department of Clinical and Biological Sciences, University of Turin
Locations (5):
- Italy (5):
  - Elisabetta Nobili, Bologna, Bologna
  - Lucia Tozzi, San Giovanni Rotondo, Foggia
  - Nicola Fazio, Milan, Milan
  - Anna Ferrero, Orbassano, Turin
  - Enrica Milanesi, Turin, Turin

REFERENCES:
- [Background] Brizzi MP, Berruti A, Ferrero A, Milanesi E, Volante M, Castiglione F, Birocco N, Bombaci S, Perroni D, Ferretti B, Alabiso O, Ciuffreda L, Bertetto O, Papotti M, Dogliotti L. Continuous 5-fluorouracil infusion plus long acting octreotide in advanced well-differentiated neuroendocrine carcinomas. A phase II trial of the Piemonte oncology network. BMC Cancer. 2009 Nov 3;9:388. doi: 10.1186/1471-2407-9-388. PMID 19886987
- [Derived] Berruti A, Fazio N, Ferrero A, Brizzi MP, Volante M, Nobili E, Tozzi L, Bodei L, Torta M, D'Avolio A, Priola AM, Birocco N, Amoroso V, Biasco G, Papotti M, Dogliotti L. Bevacizumab plus octreotide and metronomic capecitabine in patients with metastatic well-to-moderately differentiated neuroendocrine tumors: the XELBEVOCT study. BMC Cancer. 2014 Mar 14;14:184. doi: 10.1186/1471-2407-14-184. PMID 24628963